CLINICAL TRIAL: NCT05820685
Title: Dronabinol On the Pain Experience (DOPE): a Pragmatic Randomized Clinical Trial
Brief Title: Dronabinol On the Pain Experience
Acronym: DOPE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study concluded because of drug shortage
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Eastern Association for the Surgery of Trauma (Unknown)
Responsible Party: Principal Investigator, John Andrew Harvin, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0499
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Standard of Care; Tramadol; Dronabinol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Drug: Standard of Care (acetaminophen +naproxen +gabapentin + as needed oxycodone or Tramadol)
- Standard of Care + Dronabinol (Experimental)
  Interventions: Drug: Standard of Care (acetaminophen +naproxen +gabapentin + as needed oxycodone or Tramadol); Drug: Dronabinol

INTERVENTIONS:
Drug: Standard of Care (acetaminophen +naproxen +gabapentin + as needed oxycodone or Tramadol) — Participants will receive acetaminophen 1000 mg every six hours, naproxen 500 mg every 12 hours, and gabapentin 300 mg every eight hours. Participants will also receive Oxycodone 5 mg or Tramadol 50 mg every six hours as needed for breakthrough pain. Providers will have the ability to adjust this pain regimen based on clinical judgement.
Drug: Dronabinol — Participants will receive Dronabinol 10 mg every 12 hours scheduled. Providers will have the ability to adjust this pain regimen based on clinical judgement.
  Arms: Standard of Care + Dronabinol

SUMMARY:
The purpose of this study is to identify the effect dronabinol has on opioid exposure when used as an adjunct to the current standard multi-modal pain regimen (MMPR)

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the floor, Surgical Intermediate Medical Unit (SIMU), Shock-Trauma ICU (STICU) at Memorial Herman Hospital-Texas Medical Center(MHH-TMC)

Exclusion Criteria:

* Pregnant
* Prisoner
* Patients placed in observation unit
* Non-acute trauma
* Admitted with primary burn injury
* Expired prior to admission
* Moribund
* Discharge from emergency department
* Left against medical advice

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Harvin, MD, FACS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Started | 241 | 243
Completed | 235 | 234
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Population: Includes all participant who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Standard of Care + Dronabinol | Total
Number analyzed (Participants) | 235 | 234 | 469
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [27 to 59] | 38 [27 to 52] | 38 [27 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 67 | 127
  Male | 175 | 167 | 342
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66 | 77 | 143
  Black | 66 | 64 | 130
  Hispanic | 83 | 83 | 166
  Other | 20 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 235 | 234 | 469
Score on Abbreviated Injury Scale (AIS) - Head [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 2]
Score on Abbreviated Injury Scale (AIS) - Chest [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 1 [0 to 3] | 2 [0 to 3] | 1 [0 to 3]
Score on Abbreviated Injury Scale (AIS) - Abdomen [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
Score on Abbreviated Injury Scale (AIS) - Extremity [Median (Inter-Quartile Range); unit: score on a scale] — The AIS classifies individual injuries by body region as follows: 0 = No Injury; 1 = Minor; 2 = Moderate; 3 = Serious; 4 = Severe; 5 = Critical; 6 = Maximal (currently untreatable)
  score on a scale | 2 [0 to 3] | 2 [0 to 3] | 2 [0 to 3]
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: score on a scale] — The Injury Severity Score (ISS) assesses the combined effects of injuries in multiple anatomical locations and ranges from from 1 to 75, with 75 being the most severe.
  score on a scale | 17 [9 to 22] | 14 [9 to 19] | 14 [9 to 21]
Number of Participants with a blunt injury [Count of Participants; unit: Participants] | 181 | 175 | 356
Number of Participants with Rib Fractures [Count of Participants; unit: Participants] | 102 | 100 | 202
Number of participants with flail segment [Count of Participants; unit: Participants] — Flail segment is the condition of having three or more contiguous ribs fractured in two or more places
  Participants | 19 | 6 | 25
Number of participants with long bone fracture [Count of Participants; unit: Participants] | 79 | 72 | 151
Number of participants with vertebral body fracture [Count of Participants; unit: Participants] | 39 | 43 | 82
Number of participants with pelvis or acetabulum fracture [Count of Participants; unit: Participants] | 49 | 37 | 86
Number of participants with traumatic brain injury [Count of Participants; unit: Participants] | 25 | 32 | 57
Number of participants who underwent laparotomy procedure [Count of Participants; unit: Participants] | 24 | 30 | 54
Number of participants who underwent thoracotomy procedure [Count of Participants; unit: Participants] | 0 | 0 | 0
Number of participants who underwent amputation procedure [Count of Participants; unit: Participants] | 7 | 3 | 10
Number of participants who underwent any procedure [Count of Participants; unit: Participants] | 181 | 184 | 365
Number of Participants With Prior Opioid Use [Count of Participants; unit: Participants]
  No | 145 | 151 | 296
  Yes | 84 | 68 | 152
  Unknown | 6 | 15 | 21
Number of Participants with a History of Smoking [Count of Participants; unit: Participants]
  No | 149 | 146 | 295
  Yes | 76 | 76 | 152
  Unknown | 10 | 12 | 22
Number of Participants with a Positive Alcohol Screen [Count of Participants; unit: Participants]
  No | 91 | 85 | 176
  Yes | 37 | 35 | 72
  Not Performed | 107 | 114 | 221
Number of Participants with a Positive Drug Screen [Count of Participants; unit: Participants]
  No | 145 | 140 | 285
  Yes | 44 | 39 | 83
  Not Performed | 46 | 55 | 101
Number of rib fractures (all participants) [Median (Inter-Quartile Range); unit: rib fractures] | 0 [0 to 4] | 0 [0 to 3] | 0 [0 to 4]
number of rib fractures (only participants with rib fractures) [Median (Inter-Quartile Range); unit: rib fractures] — Population: 102 participant in the Standard of Care arm had rib fractures. 100 participant in the Standard of Care + Dronabinol arm had rib fractures. This baseline measure is for participants with rib fractures.
  rib fractures
    number analyzed (Participants) | 102 | 100 | 202
    (all) | 5 [2 to 8] | 4 [2 to 6] | 5 [2 to 7]
Unit of admission [Count of Participants; unit: Participants]
  Floor | 164 | 167 | 331
  Intermediate unit | 32 | 31 | 63
  Intensive care unit | 32 | 33 | 65
  Other | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Milligram Equivalents (MME) Per Day
Description: This will be calculated by calculated by taking the total of MMEs from all opioids received and dividing by length of stay
Time Frame: From time of admission to time of discharge (about 11 days after admission)
Measure: Median (Inter-Quartile Range); unit: MME Per Day
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
MME Per Day | 15 [9 to 25] | 17 [10 to 26]

2. Secondary Outcome: Total Morphine Milligram Equivalents (MME) Over Hospital Stay
Description: This will be calculated by calculated by taking the total of MMEs from all opioids received
Time Frame: From time of admission to time of discharge (about 11 days after admission)
Measure: Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents (MME)
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
Morphine Milligram Equivalents (MME) | 99 [50 to 197] | 99 [48 to 182]

3. Secondary Outcome: Pain as Assessed by the Defense and Veterans Pain Rating Scale (DVPRS)
Description: This is a 4 item questionnaire and each is scored from 0(no pain) to 10( as bad as it could be, nothing else matters), enhanced with functional word descriptor anchors at each pain level and "traffic light" color coded bars to delineate levels of pain; mild (1 to 4, green), moderate (5 to 6, yellow), and severe (7 to 10, red) pain a higher number indicating more pain Average pain score during the course of the hospital stay will be reported.
Time Frame: From time of admission to time of discharge (about 11 days after admission)
Population: Data were not collected for this outcome measure because it was not charted by the bedside nurse.
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants Discharged Form Hospital With a Prescription for an Opioid Medication
Time Frame: Discharge (about 11 days after admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
Participants | 133 | 144

5. Secondary Outcome: Number of Participants Discharged Form Hospital Without a Prescription for an Opioid Medication
Time Frame: Discharge (about 11 days after admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
Participants | 102 | 90

6. Secondary Outcome: Number of Participants That Have Incidences of Opioid-related Complications, Such as Ileus, Aspiration, Unplanned Intubation, Unplanned Admission to an Intensive Care Unit, and Use of an Opioid-reversal Agent.
Time Frame: From time of admission to time of discharge (about 11 days after admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
Participants | 10 | 13

7. Secondary Outcome: Hospital Length of Stay
Time Frame: From time of admission to time of discharge (about 11 days after admission)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
days | 6 [4 to 11] | 6 [3 to 9]

8. Secondary Outcome: Number of Hospital Free Days
Description: This will be calculated as (30 days-length of stay (LOS))
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 235 | 234
Days | 24 [19 to 26] | 24 [21 to 27]

9. Secondary Outcome: ICU Length of Stay (Participants With >0 ICU Days)
Time Frame: From time of admission to ICU to time of discharge from ICU (about 12 days after admission)
Population: Only the participants with > 0 ICU days were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 39 | 42
days | 5 [3 to 12] | 6 [3 to 10]

10. Secondary Outcome: Number of Days on a Ventilator (Participants With > 0 Days on a Ventilator)
Time Frame: From time of intubation to time of extubation (about 14 days after admission)
Population: Only the participants with > 0 days on a ventilator were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 23 | 23
days | 3 [2 to 11] | 6 [3 to 14]

11. Secondary Outcome: Number of ICU Free Days (Participants With >0 ICU Days)
Description: This will be calculated as (30 days-number of days in ICU)
Time Frame: 30 days
Population: Only the participants with > 0 ICU days were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 39 | 42
days | 25 [18 to 27] | 25 [20 to 27]

12. Secondary Outcome: Number of Ventilator Free Days (Participants With >0 Days on a Ventilator)
Description: This will be calculated as (30 days-number of days spent on ventilator)
Time Frame: 30 days
Population: Only the participants with > 0 days on a ventilator were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Standard of Care + Dronabinol
Number analyzed (Participants) | 23 | 23
days | 27 [19 to 28] | 24 [16 to 27]

ADVERSE EVENTS:
Time Frame: From hospital admission up to hospital discharge (about 11 days)
Arm/Group | Standard of Care | Standard of Care + Dronabinol
All-Cause Mortality (participants affected / at risk) | 5/235 | 4/234
Serious Adverse Events (participants affected / at risk) | 10/235 | 13/234
Other Adverse Events (participants affected / at risk) | 0/235 | 0/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=235) | Standard of Care + Dronabinol (N=234)
Unplanned intubation (General disorders) | 3 | 4
Unplanned ICU (Gastrointestinal disorders) | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT05820685/Prot_SAP_000.pdf